CLINICAL TRIAL: NCT01781364
Title: Neuroplasticity-oriented Cognitive Intervention in Early Onset and First Admission Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Prof. Dr. Brigitte Rockstroh, Prof. Dr., University of Konstanz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FP16963311
Record Dates: First submitted 2013-01-22; First posted 2013-02-01 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Psychosis
Keywords: Brain Oscillations; Cognitive Performance
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive Training (Experimental): Brain Fitness Training, Posit Science SF
  Interventions: Behavioral: Brain Fitness Training, Posit Science SF

INTERVENTIONS:
Behavioral: Brain Fitness Training, Posit Science SF — Computer aided cognitive training based on principles of neuroplasticity

SUMMARY:
The purpose of this study is to reveal the specific effects of computer-aided cognitive training on course and rehabilitation in early onset schizophrenia

DETAILED DESCRIPTION:
Impairment in cognitive functions is one of the main symptoms in schizophrenia and is currently one of the challenges in the treatment of the disease. We examine the beneficial effect of computer-aided training program on course and rehabilitation of young psychotic patients with early onset psychosis. In addition we develop predictors for the course of disorder from neuroimaging data.

ELIGIBILITY:
Inclusion Criteria:

* Early Onset Psychosis

Exclusion Criteria:

* Chronicity
* Insufficient German skills

Ages: 17 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
change from baseline at post-training and at 3-months and at 7-months follow-up in each of the following outcome measures: neuropsychological test performance (MCCCB), GAF, PANSS, MEG event-related potentials (M50), alpha activity | baseline, post-training (training duration 4 weeks), 3-month follow-up, 7-month follow-up

SECONDARY OUTCOMES:
change from baseline in GAF score at 3-months and 7-moths follow-up | baseline, 3-months follow-up, 7-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte S Rockstroh, Prof. Dr., Study Director — University of Konstanz
Locations (1):
- University Konstanz, Konstanz, Baden-Wurttemberg, Germany